CLINICAL TRIAL: NCT01815697
Title: A Prospective, Randomized Study of Enhanced External Counterpulsation in Patients With Lower Urinary Tract Symptoms
Brief Title: Effect of Enhanced External Counterpulsation on Lower Urinary Tract Symptoms
Acronym: EECPLUTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Sheng Fu,MD, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSFC-81070488
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia; Urinary Retention; Vascular Endothelium; Counterpulsation, External
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Urinary Retention

STUDY DESIGN:
Intervention Model Description: Patients with benign prostatic hyperplasia are assigned to two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced External Counterpulsation (Experimental): Men with benign prostatic hyperplasia receive 35- 36 hours Enhanced External Counterpulsation treatment
  Interventions: Device: Enhanced External Counterpulsation
- Control (No Intervention): Men with benign prostatic hyperplasia without Enhanced External Counterpulsation treatment as control

INTERVENTIONS:
Device: Enhanced External Counterpulsation — Enhanced external counterpulsation (EECP) is mainly used in cardiovascular and cerebrovascular diseases, which has been proven to be able to improve microcirculation and endothelial function. EECP therapy is done by sequential inflation of 3 sets of cuffs wrapped around the lower extremities during diastole and deflation of the cuffs during systole. The systolic deflation/ Diastolic inflation sequence of EECP leads to systolic unloading and diastolic augmentation, resulting in increased blood flow in a pulsatile manner. The patients will receive 35-36 hours EECP intervention, 1-hour session every day over a 7-week period.
  Other Names: EECP
  Arms: Enhanced External Counterpulsation

SUMMARY:
The purpose of this study is to access the effects of Enhanced External Counterpulsation treatment on lower urinary tract symptoms in patients with benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Patients with benign prostatic hyperplasia and will be randomized into two groups: EECP intervention or not. Lower urinary tract symptoms, hemodynamic parameters, vascular endothelial function will be measured and compared

ELIGIBILITY:
Inclusion Criteria:

1. men over 18 years old;
2. provide signed informed consent;
3. existence of lower urinary tract symptoms
4. agree not to use any lower urinary tract symptoms treatment at least one month;
5. suitable for receiving EECP treatment

Exclusion Criteria:

1. history of long drug abuse;
2. pelvic, spine, brain trauma or surgery;
3. endocrine, liver, lung, kidney disease, malignancies, hematological disorders;
4. Severe infection without effective control；
5. lower limbs deep vein thrombosis；
6. Large area of ulcerative rash；
7. unsuitable for receiving EECP treatment

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lower urinary tract symptoms evaluated by International Prostate Symptom Score | 7 weeks

SECONDARY OUTCOMES:
Urinary flow rate | 7 weeks
  Change from baseline in urinary flow rate
Endothelial function | 7 weeks
  Change from baseline in flow- mediated dilation (FMD) accessed by color Doppler ultrasound system

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M. D., Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat- sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No